CLINICAL TRIAL: NCT04064762
Title: Targeted Plasticity Therapy for Posttraumatic Stress Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Defense Advanced Research Projects Agency (U.S. Federal Agency); The University of Texas at Dallas (Other); University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 019-280; N66001-15-2-4057 (Other Grant/Funding Number: Defense Advanced Research Projects Agency (DARPA))
Record Dates: First submitted 2019-07-31; First posted 2019-08-22 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Vagus Nerve Stimulation (VNS); Prolonged Exposure Therapy (PE); PTSD; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Vagus Nerve Stimulation + Prolonged Exposure Therapy (Experimental): Study treatment is vagus nerve stimulation (VNS) delivered during Prolonged Exposure Therapy.
  Interventions: Device: Paired Vagus Nerve Stimulation

INTERVENTIONS:
Device: Paired Vagus Nerve Stimulation — Stimulation of the vagus nerve that is paired with Prolonged Exposure Therapy.
  Other Names: VNS; vagus nerve stimulation; paired VNS

SUMMARY:
Posttraumatic stress disorder is a debilitating condition that develops in the aftermath of a traumatic experience, leading to hyperarousal, heightened anxiety, and uncontrolled fear that can be driven by intrusive memories or trauma reminders. The Texas Biomedical Device Center has developed a novel technique, termed targeted plasticity therapy (TPT), to boost neuroplasticity in conjunction with various forms of rehabilitation, including prolonged exposure therapy. The technique involves stimulation of the vagus nerve. The purpose of this open-label pilot study is to assess the safety of using a new device to deliver vagus nerve stimulation to reduce symptom severity in participants with PTSD when paired with prolonged exposure therapy. Additionally, the study will assess the prospective benefit of the system and garner an initial estimate of efficacy for a subsequent trial.

ELIGIBILITY:
Inclusion Criteria

* Patients diagnosed with chronic PTSD for at least 3 months based on the DSM-5 criteria (PSSI-5 score of 9-45)
* Appropriate candidate for VNS implantation
* Adult, aged 18-64
* Provision of signed and dated informed consent form
* Willingness to comply with all study procedures and availability for the duration of the study
* Right vocal cord has normal movement when assessed by laryngoscopy
* Women of reproductive potential must use contraceptive protection

Exclusion Criteria

* PSSI-5 score of 46 or greater (very severe symptoms)
* Current substance dependence
* Currently undergoing prolonged exposure therapy elsewhere
* Concomitant clinically significant brain injuries
* Prior injury to vagus nerve
* Prior or current treatment with vagus nerve stimulation
* Participant receiving any therapy (medication or otherwise) that would interfere with VNS
* Planning to become pregnant, currently pregnant, or lactating
* Clinical complications that hinder or contraindicate the surgical procedure
* Cognitive impairment that would interfere with study participation, confirmed by medical evaluation (will be assessed through chart review and with the Cognistat)
* Psychological conditions such as schizophrenia, bipolar disorder, or psychosis that could interfere with study participation and follow-up
* Participation in other interventional clinical trial
* Participants with known immunodeficiency including participants who are receiving or have received chronic corticosteroids, immunosuppressants, immunostimulating agents or radiation therapy within 6 months
* Significant comorbidities or conditions associated with high risk for surgical or anesthetic survival (e.g. renal failure, unstable cardiac disease, poorly controlled diabetes, immunosuppression, etc.).
* Active neoplastic disease.
* Significant local circulatory problems that would interfere with device implantation and communication, (e.g. thrombophlebitis and lymphedema).
* Any condition which, in the judgment of the Investigator, would preclude adequate evaluation of device's safety and performance.
* Incarceration or legal detention
* Non-English speaking
* Patients who are acutely suicidal and/or have been admitted for a suicide attempt

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events [Device Safety] | From Week 1 through study follow-up, approximately two years from the date of implant
  Review of adverse events reported throughout the trial will be used to inform the potential risks associated with the ReStore system and provide a better understanding of risk/benefit analysis.

SECONDARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Weeks 1, 9, 15, 19, 36, 62
  The CAPS-5 is a 30-item structured PTSD diagnostic interview that measures PTSD symptoms. (Weathers, Bovin, Lee, et al. 2018).
PTSD Checklist for DSM-5 (PCL-5) | Weeks 1, 9-15, 19, 36, 62
  The PCL-5 is a 20 item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. (Weathers, Litz, Keane, et al. 2013).
Patient Health Questionnaire-9 (PHQ-9) | Weeks 1, 9-15, 19, 36, 62
  The PHQ-9 is a brief self-report measure of major depressive disorder (Kroenke et al, 2001). The PHQ-9 is considered to be a valid measure of depression for population-based studies and clinical populations (Corson, Gerrity, & Dobscha, 2004) with a cut off score of equal or greater than 10 as the diagnostic for current depression.
Generalized Anxiety Disorder 7-item Scale (GAD-7) | Weeks 9, 15, 19, 36, 62
  The GAD7 is a 7-item questionnaire that measures severity of anxiety (Spitzer et al, 2006). Response options are "not at all," "several days," "more than half the days," and "nearly every day," scored as 0, 1, 2, and 3, respectively. Therefore, GAD-7 scores range from 0 to 21, with scores of 5, 10, and 15 representing mild, moderate, and severe anxiety symptom levels, respectively.
Posttraumatic Cognitions Inventory (PTCI) | Weeks 9-15, 19, 36, 62
  The PTCI is a 36-item instrument that assesses dysfunctional post-trauma cognitions across self, world, and self-blame to yield a total score (Foa et al., 1999). The scale has high internal consistencies (.97, .88, .86, .97, respectively) and correlates well with PTSD severity, anxiety, and depression (.44 to .79).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kilgard, PhD, Principal Investigator — The University of Texas at Dallas; Robert Rennaker, PhD, Principal Investigator — The University of Texas at Dallas; Seth Hays, PhD, Study Director — The University of Texas at Dallas; Jane Wigginton, MD, Principal Investigator — University of Texas Southwestern Medical Center; Michael Foreman, MD FACS, Principal Investigator — Baylor Health Care System; Mark Powers, PhD, Study Director — Baylor Health Care System; Richard Naftalis, MD, FAANS, FACS, Study Director — Baylor Health Care System; Ann Marie Warren, PhD, Study Director — Baylor Health Care System; Jasper Smits, PhD, Study Director — The University of Texas at Austin
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders. 5th ed. Washington, DC: American Psychiatric Association; 2013.
- [Background] Corson K, Gerrity MS, Dobscha SK. Screening for depression and suicidality in a VA primary care setting: 2 items are better than 1 item. Am J Manag Care. 2004 Nov;10(11 Pt 2):839-45. PMID 15609737
- [Background] Engineer ND, Riley JR, Seale JD, Vrana WA, Shetake JA, Sudanagunta SP, Borland MS, Kilgard MP. Reversing pathological neural activity using targeted plasticity. Nature. 2011 Feb 3;470(7332):101-4. doi: 10.1038/nature09656. Epub 2011 Jan 12. PMID 21228773
- [Background] Foa EB, Ehlers A, Clark DM, Tolin DF, Orsillo SM. The Posttraumatic Cognitions Inventory (PTCI): Development and validation. Psychol Assess 11(3): 303-314, 1999.
- [Background] Foa EB, McLean CP, Zang Y, Zhong J, Powers MB, Kauffman BY, Rauch S, Porter K, Knowles K. Psychometric properties of the Posttraumatic Diagnostic Scale for DSM-5 (PDS-5). Psychol Assess. 2016 Oct;28(10):1166-1171. doi: 10.1037/pas0000258. Epub 2015 Dec 21. PMID 26691504
- [Background] Foa EB, McLean CP, Zang Y, Zhong J, Rauch S, Porter K, Knowles K, Powers MB, Kauffman BY. Psychometric properties of the Posttraumatic Stress Disorder Symptom Scale Interview for DSM-5 (PSSI-5). Psychol Assess. 2016 Oct;28(10):1159-1165. doi: 10.1037/pas0000259. Epub 2015 Dec 21. PMID 26691507
- [Background] Gilboa-Schechtman E, Foa EB, Shafran N, Aderka IM, Powers MB, Rachamim L, Rosenbach L, Yadin E, Apter A. Prolonged exposure versus dynamic therapy for adolescent PTSD: a pilot randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2010 Oct;49(10):1034-42. doi: 10.1016/j.jaac.2010.07.014. Epub 2010 Sep 6. PMID 20855048
- [Background] Goodson J, Helstrom A, Halpern JM, Ferenschak MP, Gillihan SJ, Powers MB. Treatment of posttraumatic stress disorder in U.S. combat veterans: a meta-analytic review. Psychol Rep. 2011 Oct;109(2):573-99. doi: 10.2466/02.09.15.16.PR0.109.5.573-599. PMID 22238857
- [Background] Hays SA, Rennaker RL, Kilgard MP. Targeting plasticity with vagus nerve stimulation to treat neurological disease. Prog Brain Res. 2013;207:275-99. doi: 10.1016/B978-0-444-63327-9.00010-2. PMID 24309259
- [Background] Hembree EA, Rauch SAM, Foa EB. Beyond the manual: The insider's guide to Prolonged Exposure therapy for PTSD. Cogn Behav Pract 10(1): 22-30, 2003.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Powers MB, Halpern JM, Ferenschak MP, Gillihan SJ, Foa EB. A meta-analytic review of prolonged exposure for posttraumatic stress disorder. Clin Psychol Rev. 2010 Aug;30(6):635-41. doi: 10.1016/j.cpr.2010.04.007. Epub 2010 May 2. PMID 20546985
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Derived] Powers MB, Hays SA, Rosenfield D, Porter AL, Gallaway H, Chauvette G, Smits JAJ, Warren AM, Douglas M, Naftalis R, Wigginton JG, Foreman M, Kilgard MP, Rennaker RL. Vagus nerve stimulation therapy for treatment-resistant PTSD. Brain Stimul. 2025 May-Jun;18(3):665-675. doi: 10.1016/j.brs.2025.03.007. Epub 2025 Mar 15. PMID 40097094